CLINICAL TRIAL: NCT02647515
Title: Intravitreal Ranibizumab Injection as Adjuvant in the Treatment of Postvitrectomy Diabetic Vitreous Hemorrhage Accompanied by Neovascular Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Ningbo University (Other)
Responsible Party: Principal Investigator, Xi Shen, chief physician, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XShen
Record Dates: First submitted 2015-12-30; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Retinopathy; Glaucoma, Neovascular
MeSH Terms: conditions — Diabetic Retinopathy; Glaucoma, Neovascular | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Experimental)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab

SUMMARY:
To determine the efficacy of intravitreal ranibizumab injection as adjuvant therapy in the treatment of postvitrectomy diabetic vitreous hemorrhage (PDVH) accompanied by neovascular glaucoma (NVG) as a means of preventing recurrent vitreous hemorrhage （VH） and optimizing postoperative intraocular pressure（IOP）control.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* PDVH obscuring the disc and vessels for more than 14 days and no evidence of retinal detachment after primary vitrectomy for PDR-related complications such as nonclearing VH, macula-involving or macula-threatening tractional retinal detachment, or fibrovascular proliferation with vitreoretinal adhesions
* NVG occurred following PDVH less than 4 weeks (NVG was diagnosed when an IOP elevation of 22mmHg or more was accompanied by neovascularization of the iris and/or the anterior chamber angle)

Exclusion Criteria:

* intraoperative use of long-acting gas or silicone oil in primary vitrectomy, repeat vitrectomy after primary vitrectomy for retinal diseases other than VH, previous history of vitrectomy
* previous intravitreal injection of ranibizumab or bevacizumab in either eye
* previous intravitreal corticosteroids injection in either eye
* pregnancy or current oral contraceptive intake
* usage of clopidogrel bisulfate or coumadin
* uncontrolled hypertension and cardiac disease
* uncontrolled renal or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
vitreous hemorrhage | 12 months
intraocular pressure | 12 months

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Schachat AP, Oyakawa RT, Michels RG, Rice TA. Complications of vitreous surgery for diabetic retinopathy. II. Postoperative complications. Ophthalmology. 1983 May;90(5):522-30. doi: 10.1016/s0161-6420(83)34540-1. PMID 6192378
- [Background] Luke J, Nassar K, Luke M, Grisanti S. Ranibizumab as adjuvant in the treatment of rubeosis iridis and neovascular glaucoma--results from a prospective interventional case series. Graefes Arch Clin Exp Ophthalmol. 2013 Oct;251(10):2403-13. doi: 10.1007/s00417-013-2428-y. Epub 2013 Jul 28. PMID 23893090
- [Derived] Shen X, Chen Y, Wang Y, Yang L, Zhong Y. Intravitreal Ranibizumab Injection as an Adjuvant in the Treatment of Neovascular Glaucoma Accompanied by Vitreous Hemorrhage after Diabetic Vitrectomy. J Ophthalmol. 2016;2016:4108490. doi: 10.1155/2016/4108490. Epub 2016 May 16. PMID 27293875